CLINICAL TRIAL: NCT02704494
Title: Resveratrol's Effects in Diabetic Nephropathy
Acronym: ReDNeph
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mesbah Shams, MD, Associate professor of internal medicine and endocrinology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 93-01-49-9028
Record Dates: First submitted 2016-03-04; First posted 2016-03-10 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Diabetic Nephropathy
Keywords: Resveratrol; Diabetes mellitus; Diabetes complications; Diabetic nephropathies; Proteinuria; Albuminuria; renal insufficiency
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Diabetes Complications; Proteinuria; Albuminuria; Renal Insufficiency | interventions — Resveratrol; Losartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Resveratrol (Experimental): Resveratrol + Losartan
  Interventions: Drug: Resveratrol; Drug: Losartan
- Placebo (Placebo Comparator): Placebo + Losartan
  Interventions: Drug: Placebo; Drug: Losartan

INTERVENTIONS:
Drug: Resveratrol — Resveratrol 500mg daily
  Arms: Resveratrol
Drug: Placebo — Placebo 1 capsule daily
  Arms: Placebo
Drug: Losartan — Losartan 12.5mg daily

SUMMARY:
The aim of this study is to evaluate the safety and effects of resveratrol in treatment of diabetic nephropathy.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) is one of the most important public health burdens, and its prevalence has rapidly increased worldwide over the past decades. One of the most important complications of DM is nephropathy.

Resveratrol (3, 5, 4'-trihydroxystilbene) is a natural polyphenolic compound belongs to the large group of polyphenols found in different plant species. The richest natural source of resveratrol is Polygonum cuspidatum - a plant root extract of which have been used in oriental folk medicine. Considerable amounts of resveratrol were also found in skin of red grapes, peanuts, groundnuts, and red vine.

Resveratrol is considered to have beneficial effects on glucose tolerance and insulin sensitivity, the cardiovascular system, as it has been found to improve vasodilatation, ischaemic preconditioning, both of which seem to be the result of the activation of the endothelial NO synthase enzyme, and to inhibit both platelet aggregation and vascular smooth muscle cell proliferation. Resveratrol itself is an efficient antioxidant, as evidenced by both in vitro and in vivo studies, and, it has also been shown to improve diabetes-related impairments in animals.

We hypothesized that resveratrol may have a favorable effects on control of diabetic nephropathy. The aim of this study is to evaluate the safety and effects of resveratrol in treatment of diabetic nephropathy.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (DM)
* Controlled blood sugar [fasting blood sugar (FBS) <130mg/dl and glycosylated hemoglobin (A1C)<7%
* Urine albumin >20mg/lit in two separate occasions during the last 3 months period
* Serum creatinin < or = 2mg/dl

Exclusion Criteria:

* Pregnancy
* Lactation
* Alcoholism
* Liver failure (acute or chronic)
* Renal failure: serum creatinin >2mg/dl
* Glomerulonephritis
* Uncontrolled hypertension
* Congestive heart failure
* Prostate disease
* Malignancy
* Bilateral renal artery stenosis
* Any systemic disease other than DM
* Any infection or rheumatologic disorder
* Use of warfarin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Urine albumin level | 3 months
Serum creatinin | 3 months

SECONDARY OUTCOMES:
Fasting blood sugar (FBS) | 3 months
Glycosylated hemoglobin (A1C) | 3 months
Liver aminotransferases (ALT and AST) | 3 months
Serum insulin level | 3 months
Number of patients with adverse events | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Gholamhossein Ranjbar Omrani, MD, Study Chair — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Jamshid Roozbeh, MD, Principal Investigator — Shiraz Nephrology and Urology Research Center, Shiraz University of Medical Sciences; Azar Sattarinejad, MD, Principal Investigator — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences; Mesbah Shams, MD, Principal Investigator — Endocrine and Metabolism Research Center, Shiraz University of Medical Sciences
Locations (1):
- Shahid Motahhari Clinic, Shiraz University of Medical Sciences, Shiraz, Fars, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Sattarinezhad A, Roozbeh J, Shirazi Yeganeh B, Omrani GR, Shams M. Resveratrol reduces albuminuria in diabetic nephropathy: A randomized double-blind placebo-controlled clinical trial. Diabetes Metab. 2019 Jan;45(1):53-59. doi: 10.1016/j.diabet.2018.05.010. Epub 2018 Jun 8. PMID 29983230